CLINICAL TRIAL: NCT06069180
Title: To Evaluate Different Conditioning Regimens for HLA Matched Donor Transplantation in Severe Aplastic Anemia: a Prospective, Multicenter, Randomized Controlled Study
Brief Title: The Optimization of Conditioning Regimen for HLA Matched HSCT in SAA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023PHB232-001
Record Dates: First submitted 2023-10-01; First posted 2023-10-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Severe Aplastic Anemia
Keywords: HLA matched donor transplantation
MeSH Terms: conditions — Anemia, Aplastic | interventions — Busulfan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Busulfan included group (Experimental): The conditioning regimens were Bu/Flu/Cy/ATG or Bu/Cy/ATG, depending on the patient's risk factors of regimen related cardiotoxicity.
  Interventions: Drug: Busulfan
- Control group (Other): The conditioning regimens were Flu/Cy/ATG or Cy/ATG, depending on the patient's risk factors of regimen related cardiotoxicity.
  Interventions: Drug: Flu/Cy/ATG or Cy/ATG

INTERVENTIONS:
Drug: Busulfan — Conditioning regimens were Bu/Flu/Cy/ATG or Bu/Cy/ATG, depending on the patient's risk factors of regimen related cardiotoxicity.
  Arms: Busulfan included group
Drug: Flu/Cy/ATG or Cy/ATG — Conditioning regimens were Flu/Cy/ATG or Cy/ATG, depending on the patient's risk factors of regimen related cardiotoxicity.
  Arms: Control group

SUMMARY:
Hematopoietic stem cell transplantation (HSCT) from a human leukocyte antigen (HLA) -matched donor is an effective option for severe aplastic anemia (SAA), but there is no standardized and recommended conditioning regimen. The occurrence of mixed chimerism after transplantation is associated with secondary graft failure and poor failure-free survival. Previous studies have shown that Fludarabine (Flu)/ Cyclophosphamide (Cy)/ antithymocyte globulin (antithymocyte globulin), ATG) and Cy/ATG conditioning regimens had higher rates of mixed chimerism and poorer failure-free survival. A small cohort study has suggested that adding busulfan to Flu/Cy/ATG or Cy/ATG can reduce the incidence of mixed chimerism and improve failure-free survival. This study was a prospective, multicenter, randomized controlled trial to compare the efficacy and safety of different conditioning regimens in the treatment of severe aplastic anemia (SAA) after hematopoietic stem cell transplantation (HSCT) from HLA-identical sibling or unrelated donor.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as SAA/vSAA
2. Indication for hematopoietic stem cell transplantation
3. Available HLA matched sibling or unrelated donor
4. No active infection
5. No serious organ damage: liver and kidney function (ALT and AST < 2.5 times normal value, normal renal function, no cardiac insufficiency)
6. Signed informed consent
7. High risk factors of mixed chimerism, at least one of the following

   1. Age < 18 years old
   2. Ferritin level ≥2500ng/ml before transplantation

Exclusion Criteria:

1. Age > 50 years old
2. ECOG≥3
3. Active infections that were difficult to control
4. Severe liver and kidney dysfunction
5. Mental illness
6. Not signing the informed consent
7. pregnant or lactating women
8. Any condition considered by the investigators to be unsuitable for enrollment

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Failure free survival | 1 year post HSCT
  Failure free survival was defined as survival with a response to therapy.

SECONDARY OUTCOMES:
The incidence of mixed chimerism | 1 year post HSCT
  The mixed chimerism was defined as the presence of 5%-95% donor haematopoietic cells.
Regimen related toxicity | 100 days post HSCT
  The regimen related toxicity (RTT) was measured according to the Seattle Toxicity Criteria (Bearman et al, 1988).
Myeloid and platelet engraftment | 100 days post HSCT
  Myeloid and platelet engraftment were defined as international criteria.
The incidence of graft versus host disease | 100 days post HSCT for aGvHD and 1 year post HSCT for cGvHD
  The severity of acute and chronic GVHD was evaluated according to standard criteria.
The incidence of CMV and EBV reactivation | 100 days post HSCT
  The incidence of CMV and EBV reactivation was defined as CMV and EBV viremia.
The incidence of Transplantation related mortality | 1 year post HSCT
  Transplantation related mortality was defined as death without disease progression.
The probability of Overall survival | 1 year post HSCT
  Overall survival was defined as the time from transplantation to death from any cause or to the last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Deparment of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No